CLINICAL TRIAL: NCT05974826
Title: Impact of a Healthy City Preventive Program on Cardiovascular Health and Well-being: a Quasi-Experimental Controlled Longitudinal Community-Based Study (Healthy Communities 2030)
Brief Title: Healthy Communities: a Healthy City Preventive Program on Cardiovascular Health and Well-being (HC)
Acronym: HC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Science, Health and Education, Spain (Other)
Collaborators: La Caixa Foundation (Other); Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHE-003-HC
Record Dates: First submitted 2023-03-08; First posted 2023-08-03 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Heart Disease Risk Factors; Healthy Lifestyle; Health Behavior
Keywords: Healthy Lifestyle; Community health promotion; Peer-group; School-based intervention
MeSH Terms: conditions — Health Behavior | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community Intervention (town: Cardona) (Experimental): The interventions aim to encourage a healthy lifestyle, including diet education, physical activity, and wellbeing.
  The SI! Program for Secondary Schools: a four-year specially designed educational program for adolescents is applied.
  The Fifty-Fifty Program implies two stages: 1) Training period; 2) a Peer-group intervention, designed to make the subjects participate actively in their healthcare
  Interventions: Behavioral: the SI! Program for Secondary Schools (NCT03504059); Behavioral: the Fifty-Fifty Program (NCT02367963)
- Community Control (town: Sallent) (No Intervention): The participants on the control group only receive general health recommendation at the end of each assessment.

INTERVENTIONS:
Behavioral: the SI! Program for Secondary Schools (NCT03504059) — The SI! Program is implemented from 1st to 4th grade of Secondary Schools. A total of 12 hours of classroom intervention per academic year, organized through three educational units, and with active and participative methodologies, and complementary intervention in the family setting, at school and on teachers.
  Arms: Community Intervention (town: Cardona)
Behavioral: the Fifty-Fifty Program (NCT02367963) — 1. Training stage: the focus is on improving individual health, through workshops (given in person by experts), and on the challenges of changing habits supervised and supported by the SHE Foundation
  2. Peer-to-peer support group sessions: It is designed to make the subjects participate actively in their healthcare. Along the sessions subjects propose assumable health goals. Participants will be able to view videos with key messages from the workshops to continue the sustainability of the changes made, and the development of new ones. Peer-to-peer support group sessions have two phases: a) leaders will receive support from the Foundation; b) participants will become agents of change with the people around them, and also in their municipality with specific actions to promote health. The role of Foundation's will only be to monitor and resolve possible doubts.
  Arms: Community Intervention (town: Cardona)

SUMMARY:
Healthy Communities is a multidisciplinary health-promotion initiative. The objective of the present study is to determine whether such an intervention will be efficacious to improve cardiovascular health compared to the current approach.

A quasi-experimental controlled longitudinal community-based intervention study will be carried out comprising approximately 2000 individuals from the age of 12 years from the cities of Cardona (intervention city) and Sallent (control city), in Spain. The core of the intervention will be based on the previous health promotion programs developed and evaluated by the Science, Health and Education (SHE) Foundation: the SI! Program (Salud Integral -Comprehensive Health) for children, and the Fifty-Fifty Program for adults. Coupled to infrastructure development, we will promote the understanding of the benefits of active living to increase awareness on the relevance of healthy lifestyle to improve health and wellbeing in three consecutive phases (Phase 1- full supervised program; Phase 2- transition period, and Phase 3- self-community driven program), which will provide full empowerment to the community.

The primary outcome will be measured with the validated composite Fuster-BEWAT (Blood pressure, Exercise/physical activity, body Weight/BMI, Alimentation/diet, and Tobbaco/smoking) score consisting of a 0-15 scale for behaviors/health risk factors. Assessments will be performed at baseline, at 2.5 and 5 years. Follow-up assessments will be conducted to determine the between group differences (intervention vs. control) in the change of the Fuster-BEWAT score at phase 2 and phase 3.

DETAILED DESCRIPTION:
Healthy Communities is a multidisciplinary health-promotion initiative aiming to improve the health and wellbeing of individuals using an innovative combination of programs and urban design to build up a "culture of health". The main aim is to turn cities and towns into places where individuals, families, and communities can increase their health and welfare potential, and where working toward cardiovascular health and wellbeing is everyone's business.

The objective of the present study is to determine whether such an intervention will be efficacious compared to the current approach.

The hypothesize is that a healthy city will impact positively to their inhabitants by improving cardiovascular health and physical activity indices, mental health, and wellbeing. For such a purpose, a controlled longitudinal community-based intervention study will be carried out on 2000 participants (1000 in the intervention and 1000 in the control towns) 12 years or older over a period of 5 years.

The core of the intervention will be based on the previous health promotion programs developed and evaluated by the Science, Health and Education (SHE) Foundation: the SI! Program for children, and the "Fifty-Fifty" Program for adults. The effect of these interventions was proven through randomized trials and the results were published in high-impact journals (Journal of the American College of Cardiology, American Heart Journal, American Journal of Medicine, etc.).

* The "SI!" Program is a school-based intervention aimed at promoting cardiovascular Health among children aged 3 to 16 years using their proximal environment (school, teachers, and families). The intervention is designed to instill and develop healthy behaviors in relation to diet, physical activity, and emotions, all connected to cardiovascular health.
* The "Fifty-Fifty" Program is a peer-group based intervention about topics related to physical activity, nutrition, and psychological aspects of lifestyle change, which is adapted to 3 different aged groups: "Fifty-Action" for young adults aged 17 to 24 years, "Fifty-Fifty" for people aged 25 to 50 years and "Fifty-Plus" for people over 51 years of age.

Coupled to infrastructure development, we will promote the understanding of the benefits of active living to increase awareness on the relevance of healthy lifestyle to improve health and wellbeing in three consecutive phases, which will provide full empowerment to the community.

During the first phase, a full educational and behavioral change program with specific actions and activities to engage and promote health and wellbeing in the community will be implemented; while the second phase will be a transition period where the Cardona inhabitants will progressively acquire a key role in such implementation under moderate supervision. Finally, during phase 3, we expect that the community will become totally empowered to drive their own health and wellbeing promotion program under minimal supervision. A non-intervention town -Sallent, in the same area- will serve as control group.

The primary outcome will be measured with the validated composite Fuster-BEWAT score consisting of a 0-15 scale for behaviors/health risk factors related to Blood pressure, Exercise, Weight, Alimentation (diet), and Tobacco (smoking). Assessments will be performed at baseline, at 2.5 and 5 years. Follow-up assessments will be used to calculate the between group differences (intervention vs. control) for the change in the Fuster-BEWAT score at midpoint of phase 2 (after the full supervised program and during the transition period), and at phase 3 (self-community driven program). Each study visit will include clinical interview, physical examination (height, weight, waist circumference, blood pressure and heart rate), point-of-care testing of lipid and glucose profile, lifestyle and behavior questionnaires, assessment of physical activity, evaluation of muscle strength and muscle quality, and assessment of psychosocial well-being. Trained health personnel will conduct all interviews and measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 12 years
* Registered in the local census of the selected towns (Cardona or Sallent)

Exclusion Criteria:

* Age less than 12 years
* Residency out of the selected towns (Cardona or Sallent)
* Unable/unwilling to provide informed consent
* Severe diseases

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — In order to try to equate groups in a quasi-experimental design, a normative age range- and sex- group equivalence matching approach will be used to select a comparison group that has approximately equivalent characteristics to the treatment group
  The recruitment will be stratified by sex and age-groups and a minimum of 75 and a maximum of 100 individuals in each strata will be recruited.
Enrollment: 2000 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Changes of the Fuster-BEWAT | baseline, 3 and 5 years
  The primary outcome will be the change from baseline in composite Fuster-BEWAT score consisting of a 0-15 scale for the following behaviors/health risk factors (higher scores correspond to healthier lifestyles): Blood pressure (systolic and diastolic blood pressure), Exercise (minutes of vigorous and moderate physical activity), Weight (body mass index calculated as body weight divided by height squared (kg/m2), Alimentation (diet) (fruits and vegetables consumption), and Tobacco (smoking) (smoking status and number of cigarettes) (0-3 points for each domain). Higher scores correspond to healthier lifestyle behaviors. The primary outcome is whether individuals belonging to a lifestyle intervention program (intervention group) demonstrate an improvement of health related behaviors and biological parameters compared to the self-management approach (control group).

SECONDARY OUTCOMES:
Changes at follow-up visits of individual domains of the Fuster-BEWAT score | baseline, 3 and 5 years
  Mean score and change at follow-up visits for each of the individual domains assimilated in the composite Fuster-BEWAT score (0-3 points for each domain, higher scores correspond to healthier lifestyles): Blood pressure (systolic and diastolic blood pressure), Exercise (minutes of vigorous and moderate physical activity), Weight (body mass index calculated as body weight divided by height squared (kg/m2)), Alimentation (diet) (fruits and vegetables consumption), and Tobacco (smoking) (smoking status and number of cigarettes). Higher scores correspond to higher compliance to lifestyle guidelines.

OTHER OUTCOMES:
Changes at follow-up visits of blood pressure | baseline, 3 and 5 years
  Mean and change in blood pressure (systolic and diastolic) (mmHg) as assessed with a fully automated blood pressure monitor (OMRON M6 monitor).
Changes at follow-up visits of physical activity | baseline, 3 and 5 years
  Mean and change in physical activity as evaluated by self-reported the short version of the Minnesota Leisure Time Physical Activity Questionnaire (REGICOR). The questionnaire calculates energy expenditure from total physical activity, and from light, moderate and vigorous physical activity (minutes per week).
Changes at follow-up visits of body mass index | baseline, 3 and 5 years
  Mean and change in body mass index (kg/m2). Body height as measured using a stadiometer (Seca 213). Body weight as measured using the OMRON BF511 electronic scale.
Changes at follow-up visits of Mediterranean diet adherence | baseline, 3 and 5 years
  Change in the adherence to a Mediterranean diet as evaluated by a self-reported the Short Diet Quality Screener (SDQS) questionnaire. Score range=0-36 (higher scores correspond to highest healthy diet).
Changes at follow-up visits of smoking status | baseline, 3 and 5 years
  Mean and change in smoking status as evaluated by self-reported the average number of cigarettes products consumed daily.
Changes at follow-up visits of blood glucose and lipid profile | baseline, 3 and 5 years
  Mean total, LDL- and HDL-cholesterol (mg/dL), and blood glucose (mg/dL) and change at follow-up visits as evaluated by point-of-care testing. Blood glucose and lipid profile were measured using a CardioCheck Plus device and PTS-Panels test strips in capillary blood sampled with a lancet in fasting status.
Changes at follow-up visits of body fat composition | baseline, 3 and 5 years
  Mean and change in body fat mass and body lean mass as measured by bioelectrical impedance.
Changes at follow-up visits of muscle strength | baseline, 3 and 5 years
  Mean and change in muscle strength evaluated by the hand-grip test (kg)
Changes at follow-up visits of psychosocial wellbeing | baseline, 3 and 5 years
  Change in psychosocial wellbeing as evaluated by self-reported questionnaire about perceived happiness (Pemberton Happiness Index), Score range=0-10 (higher scores correspond to highest psychosocial wellbeing).
Changes at follow-up visits of perceived stress | baseline, 3 and 5 years
  Change in perceived stress as evaluated by self-reported questionnaire Perceived Stress Scale (14-items PSS). Score range=0-56 (higher scores correspond to highest perceived stress).
Changes at follow-up visits of social support | baseline, 3 and 5 years
  Change in social support as evaluated by self-reported questionnaire Spanish-translated ENRICHD Social Support Instrument. Score range=0-21 (higher scores correspond to highest social support).
Changes at follow-up visits of resilience | baseline, 3 and 5 years
  Change in resilience as evaluated by self-reported questionnaire Spanish-adaptation of Brief Resilience Coping Scale. Score range=4-20 (higher scores correspond to highest resilience).
Changes at follow-up visits of self-esteem | baseline, 3 and 5 years
  Change in self-esteem as evaluated by self-reported questionnaire Child Health and Illness Profile-Adolescent Edition (CHIP-AE). Score range=1-20 (higher scores correspond to highest self-esteem).
Changes at follow-up visits of mood | baseline, 3 and 5 years
  Change in mood as evaluated by self-reported a Spanish questionnaire design by Vazquez-Fernandez ME et al 2013. Score range=0-6 (scoring ≥3 means mood is negative).
Changes in the proportion of participants with any positive modifications in behavior | baseline, 3 and 5 years
  Changes in the proportion of participants with any positive modifications in behavior

CONTACTS AND LOCATIONS:
Overall Officials: Valentín Fuster, Principal Investigator — Mount Sinaí Hospital
Locations (1):
- Foundation for Science, Health and Education, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data underlying results in a publication will be shared on reasonable request to the principal investigator.
Time Frame: Starting 9 months after publication
Access Criteria: the de-identified data underlying results in a publication will be shared on reasonable request to the principal investigator.
  Email: estudio@fundacionshe.org
URL: https://fundacionshe.org/healthycommunities2030/

REFERENCES:
- [Background] Fernandez-Jimenez R, Santos-Beneit G, Tresserra-Rimbau A, Bodega P, de Miguel M, de Cos-Gandoy A, Rodriguez C, Carral V, Orrit X, Haro D, Carvajal I, Ibanez B, Storniolo C, Domenech M, Estruch R, Fernandez-Alvira JM, Lamuela-Raventos RM, Fuster V. Rationale and design of the school-based SI! Program to face obesity and promote health among Spanish adolescents: A cluster-randomized controlled trial. Am Heart J. 2019 Sep;215:27-40. doi: 10.1016/j.ahj.2019.03.014. Epub 2019 Apr 10. PMID 31277052
- [Background] Fernandez-Alvira JM, Fuster V, Pocock S, Sanz J, Fernandez-Friera L, Laclaustra M, Fernandez-Jimenez R, Mendiguren J, Fernandez-Ortiz A, Ibanez B, Bueno H. Predicting Subclinical Atherosclerosis in Low-Risk Individuals: Ideal Cardiovascular Health Score and Fuster-BEWAT Score. J Am Coll Cardiol. 2017 Nov 14;70(20):2463-2473. doi: 10.1016/j.jacc.2017.09.032. PMID 29145946
- [Background] Gomez-Pardo E, Fernandez-Alvira JM, Vilanova M, Haro D, Martinez R, Carvajal I, Carral V, Rodriguez C, de Miguel M, Bodega P, Santos-Beneit G, Penalvo JL, Marina I, Perez-Farinos N, Dal Re M, Villar C, Robledo T, Vedanthan R, Bansilal S, Fuster V. A Comprehensive Lifestyle Peer Group-Based Intervention on Cardiovascular Risk Factors: The Randomized Controlled Fifty-Fifty Program. J Am Coll Cardiol. 2016 Feb 9;67(5):476-85. doi: 10.1016/j.jacc.2015.10.033. Epub 2015 Nov 9. PMID 26562047
- See also: Web of the SHE Foundation — https://fundacionshe.org/
- See also: web of the Healthy Communities Program — https://fundacionshe.org/healthycommunities2030/